CLINICAL TRIAL: NCT06454110
Title: A Phase II, Open-Label Study of NM8074 in Patients With Immunoglobulin A Nephropathy (IgAN)
Brief Title: Study of NM8074 in Patients With Immunoglobulin A Nephropathy (IgAN)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NovelMed Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NM8074-IGAN-601
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: The study will enroll a planned total of 10 patients as subjects for the trial, with extra enrollment if needed, at the discretion of the Investigator. All subjects will be administered 17 mg/kg of NM8074 intravenously every week, for a total of 15 doses from Day 1 to Day 99 of the Treatment Period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): All subjects will be administered 17 mg/kg of NM8074 intravenously every week, for a total of 15 doses from Day 1 to Day 99 of the Treatment Period.
  Interventions: Drug: NM8074

INTERVENTIONS:
Drug: NM8074 — NM8074 will be administered as an intravenous infusion. All subjects will be administered 17 mg/kg of NM8074 intravenously weekly for a total of 15 doses from Day 1 to Day 99 of the Treatment Period.

SUMMARY:
This is a Phase II, open-label study designed to To evaluate the safety and efficacy of NM8074 in reducing proteinuria relative to baseline in IgAN patients after 99 days of treatment.

DETAILED DESCRIPTION:
The proposed study, NM8074-IgAN-601, will enroll a planned total of 10 patients as subjects for the trial. All subjects will be administered 17 mg/kg of NM8074 intravenously every week, for a total of 15 doses from Day 1 to Day 99 of the Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age at the time of consent.
* A body mass index (BMI) within the range of 15 - 38 kg/m2. BMI = Body weight (kg) / [Height (m)]2.
* Confirmation of IgA Nephropathy verified by biopsy performed within the previous three years.
* All patients must be vaccinated prior to dosing with MenACWY Menactra® polysaccharide diphtheria toxoid conjugate vaccination against Neisseria meningitidis serogroups A, C, Y, and W-135. MenB meningococcal serogroup B vaccine (Bexsero®) will be administered per local guidelines.
* Hemoglobin ≥ 10g/dL and platelet count ≥ 100,000/mm3
* Female and male participates must agree to use contraceptives

Exclusion Criteria:

* Evidence of severe urinary obstruction or difficulty in voiding; any urinary tract disorder other than IgAN at screening and before dosing with NM8074.
* Require dialysis or plasma exchange within 12 weeks prior to screening.
* Presence of crescent formation in ≥50% of glomeruli assessed on renal biopsy.
* History of bone marrow, hematopoietic stem cells, or solid organ transplantation.
* Use of other investigational drugs at the time of enrolment, or within 5 half-lives of enrolment or within 3 months to study day 1 whichever is longer.
* Severe concurrent co-morbidities not amenable to active treatment, e.g., patients with severe kidney disease (CKD stage 4, chronic dialysis).
* Clinically significant abnormal ECG during screening.
* Currently active systemic infection or suspicion of active bacterial, viral, or fungal infection within 2 weeks prior to first dose, or history of unexplained, recurrent bacterial infections.
* Has a currently active or known history of meningococcal disease or N. meningitidis infection.
* Clinically significant medical or psychological conditions or risk factors that, as per the Investigator's judgment, could hinder the patient's participation in the study, introduce additional risks for the patient, or complicate the evaluation of the patient or study outcomes.
* Pregnant, planning to become pregnant, or nursing female subjects.
* Females with a positive pregnancy test result at Screening or on Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline or Percent Change from Baseline in urine protein to creatinine concentration ratio | Up to Study Day 99

SECONDARY OUTCOMES:
Change from Baseline or Percent Change from Baseline in eGFR | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in Serum Creatinine | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in Hematuria | Up to Study Day 155
  Measured through red blood cells present in urine from urinalysis
Change from Baseline or Percent Change from Baseline in Urine Albumin to Creatinine concentration ratio | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in Bb plasma levels | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in sC5b-9 plasma levels | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in UPCR | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in Tmax | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in Cmax | Up to study Day 155
Change from Baseline or Percent Change from Baseline AUC0-t | Up to study Day 155
Change from Baseline or Percent Change from Baseline in CLr | Up to study Day 155
Change from Baseline or Percent Change from Baseline in quality of life (QoL) Assessed via the Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale, Version 4. | Up to study Day 155
  The FACIT-fatigue scale is a 13-item patient-reported measure of fatigue with a 7-day recall period. Items are scored on a 0 - 4 response scale ranging from "Not at all" to "Very much so". All items are summed to create a single fatigue score with a range from 0 to 52 with a better quality of life indicated by a higher score.
Change from Baseline or Percent Change from Baseline in Quality of Life (QoL) Assessed via the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 Scale (QLQ- C30), Version 3.0 | Up to study Day 155
  All EORTC QLQ-C30 scales and single-item measures range from 0 to 100. This includes 3 symptom scales (fatigue, pain, nausea and vomiting), 5 functional scales (physical, role, cognitive, emotional, and social), single-item questions addressing symptoms like insomnia, dyspnea, loss of appetite, and others that are commonly reported by cancer patients, and the perceived financial impact of the disease. A higher score is associated with a greater quality of life for global health status

OTHER OUTCOMES:
Change from Baseline or Percent Change from Baseline in Classical Pathway (CP) modulation | Up to Study Day 155
  NM8074-mediated CP inhibition is measure via a complement CP ELISA-based assay measuring MAC formation.
Change from Baseline or Percent Change from Baseline in Factor B levels | Up to Study Day 155
Change from Baseline or Percent Change from Baseline in plasma concentration of NM8074 | Up to Study Day 155
Maximum plasma concentration (Cmax) | Up to Study Day 155
Time corresponding to Cmax (tmax) | Up to Study Day 155
Area under the drug concentration-time curves (AUC0-t) | Up to Study Day 155

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SJ, Koo HM, Lim BJ, Oh HJ, Yoo DE, Shin DH, Lee MJ, Doh FM, Park JT, Yoo TH, Kang SW, Choi KH, Jeong HJ, Han SH. Decreased circulating C3 levels and mesangial C3 deposition predict renal outcome in patients with IgA nephropathy. PLoS One. 2012;7(7):e40495. doi: 10.1371/journal.pone.0040495. Epub 2012 Jul 6. PMID 22792353
- [Background] Lafayette RA, Kelepouris E. Immunoglobulin A Nephropathy: Advances in Understanding of Pathogenesis and Treatment. Am J Nephrol. 2018;47 Suppl 1:43-52. doi: 10.1159/000481636. Epub 2018 May 31. PMID 29852501
- [Background] Duval A, Caillard S, Fremeaux-Bacchi V. The complement system in IgAN: mechanistic context for therapeutic opportunities. Nephrol Dial Transplant. 2023 Nov 30;38(12):2685-2693. doi: 10.1093/ndt/gfad140. PMID 37385820
- [Background] Medjeral-Thomas NR, Cook HT, Pickering MC. Complement activation in IgA nephropathy. Semin Immunopathol. 2021 Oct;43(5):679-690. doi: 10.1007/s00281-021-00882-9. Epub 2021 Aug 11. PMID 34379175
- [Background] Stefan G, Jullien P, Masson I, Alamartine E, Mariat C, Maillard N. Circulating alternative pathway complement cleavage factor Bb is associated with vascular lesions and outcomes in IgA nephropathy. Nephrol Dial Transplant. 2023 Nov 8;38(Suppl 2):ii11-ii18. doi: 10.1093/ndt/gfad163. PMID 37816675